CLINICAL TRIAL: NCT03317249
Title: Pregnancy Related Inappropriate Sinus Tachycardia Syndrome Study
Brief Title: Pregnancy Related Inappropriate Sinus Tachycardia
Acronym: PRIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Mark Belham, Consultant Cardiologist, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: PRIST
Record Dates: First submitted 2017-10-06; First posted 2017-10-23 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Inappropriate Sinus Tachycardia; Pregnancy Related
Keywords: Inappropriate Sinus Tachycardia; Pregnancy Related; IST
MeSH Terms: interventions — Electrocardiography; Heart Rate Determination; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Healthy: Pregnant females aged between 18-45 years who do not have IST syndrome
  Interventions: Diagnostic Test: ECG; Diagnostic Test: heart rate monitor; Diagnostic Test: Autonomic Nervous System (ANS) Activity; Diagnostic Test: Haemodynamic variables; Other: Echocardiogram
- Pregnant IST: Pregnant females aged between 18-45 years who have IST syndrome
  Interventions: Diagnostic Test: ECG; Diagnostic Test: heart rate monitor; Diagnostic Test: Autonomic Nervous System (ANS) Activity; Diagnostic Test: Haemodynamic variables

INTERVENTIONS:
Diagnostic Test: ECG — 12-lead electrocardiogram
Diagnostic Test: heart rate monitor — 24-hour heart rate monitor used to calculate mean heart rate and heart rate variability
Diagnostic Test: Autonomic Nervous System (ANS) Activity — Heart Rate Variability (HRV) and Baroreflex sensitivity (BRS):
  Resting and exercise HRV and BRS calculated from ECG, Dundee Step test and blood pressure measurements.
Diagnostic Test: Haemodynamic variables — Cardiac output (CO), stroke volume (SV) and systematic vascular resistance (SVR) will be assessed and calculated using a non-invasive, inert gas re-breathing technique whereby expired gases will be sampled and analysed alongside and blood pressure measurements.
Other: Echocardiogram — optional (for non-IST participants only)
  Groups: Pregnant Healthy

SUMMARY:
A feasibility study into the exploration of possible mechanisms underlying inappropriate sinus tachycardia (IST) syndrome in pregnancy.

DETAILED DESCRIPTION:
This is a non-interventional, physiological study which will explore the feasibility of examining autonomic function and related haemodynamic variables in pregnant women with and without inappropriate sinus tachycardia, with the aim of providing scope for future research.

Sinus tachycardia (normal heart rhythm but fast heart rate) is common and usually related to an obvious cause (e.g. exercise such a running or cycling) and doesn't cause any untoward symptoms. In rare cases however, sinus tachycardia can occur without an obvious cause (i.e. it is inappropriate to the situation) and can cause distressing symptoms such as palpitations, dizziness and breathlessness at rest or with minimal exertion. This syndrome of inappropriate sinus tachycardia is poorly understood and can be difficult to manage; especially when the affected individual is pregnant. In order to understand the condition better and improve care pathways we aim to measure various features of the cardiovascular system in pregnant women with and without IST.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years of age
* Able to give written informed consent and willing to participate
* The participant falls into one of the below categories:

  i. Pregnant women with IST ii. Pregnant women without IST

Exclusion Criteria:

* Obesity (BMI > 29.9)
* Current or recent (within last 3 months) smoker
* Known medical condition likely to affect HRV (other than IST in relevant groups)
* Previous history of hypertensive disorders in pregnancy
* Lack of written informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hospital clinics (cardiology clinics and antenatal clinics)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-10-06 (Estimated); Study Completion 2020-10-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of examining autonomic function and related haemodynamic variables in pregnant women with and without inappropriate sinus tachycardia | Up to 3 years
  Number of women in each group who agree to participate in the study
Assessment of autonomic function and related haemodynamic variables in pregnant women with and without inappropriate sinus tachycardia | Up to 3 years
  Heart rate variability (HRV) at rest using time and frequency domain (e.g. SDNN ms and LF and HF), combined to give absolute power in ms².
Assessment of autonomic function and related haemodynamic variables in pregnant women with and without inappropriate sinus tachycardia | Up to 3 years
  Baroreflex sensitivity (BRS) at rest calculated from the change in systolic pressure and change in R-R interval to give change in pressure per change in RR interval, measured in milliseconds (mmHg/ms)

SECONDARY OUTCOMES:
Assessment of ANS function in pregnant women with and without IST, at rest and during mild exercise | Up to 3 years
  Stroke volume in ml
Assessment of ANS function in pregnant women with and without IST, at rest and during mild exercise | Up to 3 years
  Heart Rate Variability during mild exercise (3 minute step test) using time and frequency domain (e.g. SDNN ms and LF and HF), combined to give absolute power in ms².
Assessment of ANS function in pregnant women with and without IST, at rest and during mild exercise | Up to 3 years
  Cardiac Output in litres/minute
Assessment of ANS function in pregnant women with and without IST, at rest and during mild exercise | Up to 3 years
  Blood Pressure in mm/Hg

CONTACTS AND LOCATIONS:
Overall Officials: Mark Belham, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No